CLINICAL TRIAL: NCT06637202
Title: SB (Swedish Breast Cancer Group) 91:A Breast Conserving Surgery With or Without Postoperative Radiotherapy for Breast Cancer Stage 1-2 (<30 mm) pN0, M0
Brief Title: Swebcg 91:A RT. Breast Conserving Surgery With or Without Radiotherapy for Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LU 80/90
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postoperative radiotherapy (Active Comparator): Patients were treated with radiotherapy to 50 Gy in 25 fractions
  Interventions: Radiation: postoperative radiotherapy
- control (No Intervention): Patients received no further treatment after surgery

INTERVENTIONS:
Radiation: postoperative radiotherapy — 50 Gy in 25 fractions
  Arms: postoperative radiotherapy

SUMMARY:
The main goal of the trial was to analyse the value of radiotherapy after breast conserving surgery for patients with breast cancer, and to find groups of patients where the treatment could be omitted.

DETAILED DESCRIPTION:
The trial recruited patients between 1991-1996, and the primary outcome in terms of recurrences has been updated through the years since then. Tumour material has been collected in order to study prognostic and predictive factors for breast cancer patients that are treated today. Late side effects of the treatment are studied.

ELIGIBILITY:
Inclusion Criteria:

* female
* not over the age of 75 years
* operated because of stage 1-2 invasive adenocarcinoma of the breast
* radical excision of the tumour

Exclusion Criteria:

* earlier cancer except cancer in situ of the cervix or skin
* distant metastases

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1187 (Actual)
Dates: Start 1991-01-01 (Actual); Primary Completion 1996-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Loco-regional recurrence | 35 years
  Recurrence in the breast or regional lymph nodes

SECONDARY OUTCOMES:
survival | 35 years
  Does radiotherapy have an impact on survival?
Secondary malignancies | 35 years
  Does radiotherapy have an impact on secondandary malignancies?

CONTACTS AND LOCATIONS:
Overall Officials: Karlsson Per, MD, prof, Principal Investigator — Göteborg University, Västra Götaland Region; Erik Holmberg, PhD, Principal Investigator — Göteborg University; Emma Nimeus Malmström, MD, ass prof, Principal Investigator — Lund University, Region Skane; Fredrika Killander, MD, PhD, Principal Investigator — Region Skane, Lund University
Locations (1):
- Region Skane, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
This trial started in 1990

REFERENCES:
- [Result] Sjostrom M, Fyles A, Liu FF, McCready D, Shi W, Rey-McIntyre K, Chang SL, Feng FY, Speers CW, Pierce LJ, Holmberg E, Ferno M, Malmstrom P, Karlsson P. Development and Validation of a Genomic Profile for the Omission of Local Adjuvant Radiation in Breast Cancer. J Clin Oncol. 2023 Mar 10;41(8):1533-1540. doi: 10.1200/JCO.22.00655. Epub 2023 Jan 4. PMID 36599119
- [Result] Strell C, Stenmark Tullberg A, Jetne Edelmann R, Akslen LA, Malmstrom P, Ferno M, Holmberg E, Ostman A, Karlsson P. Prognostic and predictive impact of stroma cells defined by PDGFRb expression in early breast cancer: results from the randomized SweBCG91RT trial. Breast Cancer Res Treat. 2021 May;187(1):45-55. doi: 10.1007/s10549-021-06136-4. Epub 2021 Mar 4. PMID 33661437
- [Result] Sjostrom M, Chang SL, Fishbane N, Davicioni E, Zhao SG, Hartman L, Holmberg E, Feng FY, Speers CW, Pierce LJ, Malmstrom P, Ferno M, Karlsson P. Clinicogenomic Radiotherapy Classifier Predicting the Need for Intensified Locoregional Treatment After Breast-Conserving Surgery for Early-Stage Breast Cancer. J Clin Oncol. 2019 Dec 10;37(35):3340-3349. doi: 10.1200/JCO.19.00761. Epub 2019 Oct 16. PMID 31618132
- [Result] Sjostrom M, Chang SL, Fishbane N, Davicioni E, Hartman L, Holmberg E, Feng FY, Speers CW, Pierce LJ, Malmstrom P, Ferno M, Karlsson P. Comprehensive Transcriptomic Profiling Identifies Breast Cancer Patients Who May Be Spared Adjuvant Systemic Therapy. Clin Cancer Res. 2020 Jan 1;26(1):171-182. doi: 10.1158/1078-0432.CCR-19-1038. Epub 2019 Sep 26. PMID 31558478
- [Result] Stenmark Tullberg A, Sjostrom M, Tran L, Nimeus E, Killander F, Kovacs A, Lundstedt D, Holmberg E, Karlsson P. Combining histological grade, TILs, and the PD-1/PD-L1 pathway to identify immunogenic tumors and de-escalate radiotherapy in early breast cancer: a secondary analysis of a randomized clinical trial. J Immunother Cancer. 2023 May;11(5):e006618. doi: 10.1136/jitc-2022-006618. PMID 37208129
- [Result] Stenmark Tullberg A, Sjostrom M, Nimeus E, Killander F, Chang SL, Feng FY, Speers CW, Pierce LJ, Kovacs A, Lundstedt D, Holmberg E, Karlsson P. Integrating Tumor-Intrinsic and Immunologic Factors to Identify Immunogenic Breast Cancers from a Low-Risk Cohort: Results from the Randomized SweBCG91RT Trial. Clin Cancer Res. 2023 May 1;29(9):1783-1793. doi: 10.1158/1078-0432.CCR-22-2746. PMID 37071498
- [Result] Egelberg M, De Marchi T, Pekar G, Tran L, Bendahl PO, Tullberg AS, Holmberg E, Karlsson P, Farnebo M, Killander F, Nimeus E. Low levels of WRAP53 predict decreased efficacy of radiotherapy and are prognostic for local recurrence and death from breast cancer: a long-term follow-up of the SweBCG91RT randomized trial. Mol Oncol. 2023 Oct;17(10):2029-2040. doi: 10.1002/1878-0261.13426. Epub 2023 Apr 19. PMID 36975842
- [Result] Tutzauer J, Sjostrom M, Holmberg E, Karlsson P, Killander F, Leeb-Lundberg LMF, Malmstrom P, Nimeus E, Ferno M, Jogi A. Breast cancer hypoxia in relation to prognosis and benefit from radiotherapy after breast-conserving surgery in a large, randomised trial with long-term follow-up. Br J Cancer. 2022 May;126(8):1145-1156. doi: 10.1038/s41416-021-01630-4. Epub 2022 Feb 9. PMID 35140341
- [Result] Killander F, Wieslander E, Karlsson P, Holmberg E, Lundstedt D, Holmberg L, Werner L, Koul S, Haghanegi M, Kjellen E, Nilsson P, Malmstrom P. No Increased Cardiac Mortality or Morbidity of Radiation Therapy in Breast Cancer Patients After Breast-Conserving Surgery: 20-Year Follow-up of the Randomized SweBCGRT Trial. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):701-709. doi: 10.1016/j.ijrobp.2020.04.003. Epub 2020 Apr 14. PMID 32302682
- [Result] Stenmark Tullberg A, Puttonen HAJ, Sjostrom M, Holmberg E, Chang SL, Feng FY, Speers C, Pierce LJ, Lundstedt D, Killander F, Nimeus E, Kovacs A, Karlsson P. Immune Infiltrate in the Primary Tumor Predicts Effect of Adjuvant Radiotherapy in Breast Cancer; Results from the Randomized SweBCG91RT Trial. Clin Cancer Res. 2021 Feb 1;27(3):749-758. doi: 10.1158/1078-0432.CCR-20-3299. Epub 2020 Nov 4. PMID 33148672
- [Result] Sjostrom M, Veenstra C, Holmberg E, Karlsson P, Killander F, Malmstrom P, Nimeus E, Ferno M, Stal O. Expression of HGF, pMet, and pAkt is related to benefit of radiotherapy after breast-conserving surgery: a long-term follow-up of the SweBCG91-RT randomised trial. Mol Oncol. 2020 Nov;14(11):2713-2726. doi: 10.1002/1878-0261.12803. Epub 2020 Sep 28. PMID 32946618
- [Result] Killander F, Karlsson P, Anderson H, Mattsson J, Holmberg E, Lundstedt D, Holmberg L, Malmstrom P. No breast cancer subgroup can be spared postoperative radiotherapy after breast-conserving surgery. Fifteen-year results from the Swedish Breast Cancer Group randomised trial, SweBCG 91 RT. Eur J Cancer. 2016 Nov;67:57-65. doi: 10.1016/j.ejca.2016.08.001. Epub 2016 Sep 7. PMID 27614164
- [Result] Lundstedt D, Gustafsson M, Malmstrom P, Johansson KA, Alsadius D, Sundberg A, Wilderang U, Holmberg E, Anderson H, Steineck G, Karlsson P. Symptoms 10-17 years after breast cancer radiotherapy data from the randomised SWEBCG91-RT trial. Radiother Oncol. 2010 Nov;97(2):281-7. doi: 10.1016/j.radonc.2010.09.018. Epub 2010 Oct 20. PMID 20970212
- [Derived] Egelberg M, De Marchi T, Schultz N, Tran L, Karlsson P, Holmberg E, Pekar G, Killander F, Nimeus E. The potential radiosensitization target PFKFB3 is related to response to radiotherapy in SweBCG91RT: a randomized clinical trial with long-term follow-up. BMC Cancer. 2025 Feb 28;25(1):374. doi: 10.1186/s12885-025-13703-1. PMID 40022029